CLINICAL TRIAL: NCT02755116
Title: Olanzapine for the Treatment of Post-Discharge Nausea and Vomiting After Ambulatory Surgery
Brief Title: Olanzapine for Nausea After Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jaime B Hyman (Other)
Responsible Party: Sponsor-Investigator, Jaime B Hyman, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GCO 15-1297
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Results first posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Nausea; Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olanzapine (Experimental): 10mg pill
  Interventions: Drug: Olanzapine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olanzapine — 10mg of olanzapine by mouth prior to anesthetic induction
  Other Names: Zyprexa; 132539-06-1; Zyprexa Zydis; Olansek; Symbyax2-Methyl-4-(4-methyl-1-piperazinyl)-10H-thieno[2,3-b][1,5]benzodiazepine
  Arms: Olanzapine
Drug: Placebo — placebo by mouth prior to anesthetic induction
  Arms: Placebo

SUMMARY:
Ambulatory surgery is occurring with rapidly increasing frequency as surgical and anesthetic techniques have improved and pressure to reduce health-care costs has increased. While there are many benefits to recovering from surgery within the home, a significant disadvantage is the lack of rapid access to a healthcare provider when postoperative complications occur. Postoperative nausea and vomiting (PONV) are common after surgery and anesthesia, and recent studies have demonstrated a high incidence of post-discharge nausea and vomiting (PDNV) after ambulatory surgery, particularly in high-risk groups (female gender, age less than 50 years, history of PONV, opioid administration in the post-anesthesia care unit (PACU), and nausea in the PACU). Current practices known to reduce the risk of postoperative nausea and vomiting in the PACU, such as the avoidance of volatile anesthetics and the use of intraoperative ondansetron and steroids, have little effect on the risk of delayed PDNV. Novel strategies to prevent PDNV are needed. Orally administered olanzapine, which has been shown to decrease the incidence of chemotherapy-induced nausea and vomiting, demonstrates promise as a novel strategy for preventing PDNV. It has a long half-life, allowing for a single dose to be administered preoperatively. This study will evaluate whether there is a difference in the incidence and severity of PDNV between patients who receive oral olanzapine versus placebo prior to general anesthesia for ambulatory surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults age ≥ 18 and ≤ 50 years old
* Patient scheduled to undergo ambulatory surgery under general anesthesia
* Willing and able to provide informed consent

Exclusion Criteria:

* Unable to swallow pills
* Current use of typical or atypical anti-psychotic medications
* History of allergy to olanzapine
* Pregnancy/Lactation (subjects of child-bearing potential will have a urine pregnancy test performed the day of surgery)
* History of QTc > 450ms or torsades de pointes
* Current use of antihypertensive medication
* Diabetes Mellitus
* Clinically significant cardiovascular disease defined as follows:

  1. Myocardial infarction or unstable angina within 6 months prior to the day of planned surgery.
  2. History of serious ventricular arrhythmia (i.e.: ventricular tachycardia or ventricular fibrillation) or cardiac arrhythmias requiring anti-arrhythmic medications, except for atrial fibrillation that is well controlled on anti-arrhythmic medication.
  3. New York Heart Association (NYHA) Class II or higher congestive heart failure.
* Postural hypotension or vasovagal syncope within 6 months of planned surgery.
* Hypotension on day of surgery, defined as a systolic blood pressure < 90mm Hg or a diastolic pressure < 60mm Hg.
* Seizure disorder
* Clinically active prolactinoma
* Hepatic disease
* Poorly controlled diabetes
* Pre-operative blood glucose > 250 mg/dL
* Narrow angle glaucoma
* Parkinson's disease
* Lewy body dementia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2016-04; Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime B Hyman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apfel CC, Philip BK, Cakmakkaya OS, Shilling A, Shi YY, Leslie JB, Allard M, Turan A, Windle P, Odom-Forren J, Hooper VD, Radke OC, Ruiz J, Kovac A. Who is at risk for postdischarge nausea and vomiting after ambulatory surgery? Anesthesiology. 2012 Sep;117(3):475-86. doi: 10.1097/ALN.0b013e318267ef31. PMID 22846680
- [Result] Hyman JB, Park C, Lin HM, Cole B, Rosen L, Fenske SS, Barr Grzesh RL, Blank SV, Polsky SB, Hartnett M, Taub PJ, Palvia V, DeMaria S Jr, Ascher-Walsh C. Olanzapine for the Prevention of Postdischarge Nausea and Vomiting after Ambulatory Surgery: A Randomized Controlled Trial. Anesthesiology. 2020 Jun;132(6):1419-1428. doi: 10.1097/ALN.0000000000003286. PMID 32229754

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 180 patients consented, 36 excluded prior to study drug administration and 144 patients were randomized and enrolled.
Groups:
- Olanzapine: 10-mg dose of olanzapine by mouth prior to anesthetic induction
Period: Overall Study
Arm/Group | Olanzapine | Placebo
Started | 74 | 70
Completed | 71 | 69
Not Completed | 3 | 1
Not completed — surgery converted to open, pt admitted | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olanzapine | Placebo | Total
Number analyzed (Participants) | 71 | 69 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (7) | 37 (7) | 37 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 69 | 140
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 27 | 53
  Not Hispanic or Latino | 45 | 42 | 87
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 14 | 24
  White | 26 | 28 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 35 | 27 | 62
American Society of Anesthesiologists (ASA) Physical Status [Count of Participants; unit: Participants] — ASA 1: A normal healthy patient. ASA 2: A patient with a mild systemic disease. ASA 3: A patient with a severe systemic disease that is not life-threatening. ASA 4: A patient with a severe systemic disease that is a constant threat to life.
  ASA 5: A moribund patient who is not expected to survive without the operation. The patient is not expected to survive beyond the next 24 hours without surgery.
  ASA 6: A brain-dead patient whose organs are being removed with the intention of transplanting them into another patient.
  Participants
    I | 19 | 24 | 43
    II | 49 | 41 | 90
    III | 3 | 4 | 7
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.8 (6.3) | 27.7 (5.9) | 27.7 (6.1)
History of postoperative nausea/vomiting [Count of Participants; unit: Participants] | 19 | 17 | 36
Motion Sickness [Count of Participants; unit: Participants] | 21 | 25 | 46
Nonsmoker [Count of Participants; unit: Participants] | 67 | 62 | 129
Number of Risk Factors [Count of Participants; unit: Participants]
  2 | 4 | 7 | 11
  3 | 43 | 35 | 78
  4 | 24 | 27 | 51
Surgery type [Count of Participants; unit: Participants]
  Laparoscopic gynecologic | 54 | 58 | 112
  Hysteroscopy | 11 | 9 | 20
  Vaginal | 3 | 1 | 4
  Plastics | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Nausea and/or Vomiting
Description: Number of participants with post-discharge nausea and/or vomiting
Time Frame: in 24 hours after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 71 | 69
Participants | 10 | 26
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority; p = 0.003, log-binomial regression; Adjusted relative risk = 0.76, 95% CI 2-sided [0.48 to 1.20]

2. Primary Outcome: Number of Participants With Severe Nausea
Description: Number of participants with severe postdischarge nausea, defined as numerical rating scale score greater than 3. (11-point numerical rating scale from 0-10, higher score indicating worse nausea)
Time Frame: in 24 hours after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 71 | 69
Participants | 4 | 14

3. Secondary Outcome: Number of Participants With Postdischarge Vomiting
Description: Number of participants with post discharge vomiting
Time Frame: in 24 hours after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 71 | 69
Participants | 2 | 8

4. Secondary Outcome: Number of Participants With PONV
Description: Number of participants with postoperative nausea and/or vomiting (PONV) in first 24 hours
Time Frame: first 24 hours post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 71 | 69
Participants | 22 | 35

5. Secondary Outcome: Number of Participants With Severe PONV
Description: Number of participants with severe PONV in first 24 hours after post-op.defined as numerical rating scale score greater than 3. (11-point numerical rating scale from 0-10, higher score indicating worse nausea)
Time Frame: first 24 hours post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 71 | 69
Participants | 12 | 26

ADVERSE EVENTS:
Time Frame: 24 hours after discharge
Arm/Group | Olanzapine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/69
Other Adverse Events (participants affected / at risk) | 24/71 | 27/69
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olanzapine (N=71) | Placebo (N=69)
Dizziness or lightheadedness (Nervous system disorders) | 21 | 27
Visual disturbances (Eye disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/16/NCT02755116/Prot_SAP_000.pdf